CLINICAL TRIAL: NCT01341561
Title: The Relevance of Biochemical Markers in the Process of Weaning
Brief Title: Relevance of Biomarkers in the Process of Weaning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. Evangelos Giannitsis, Department of Cardiology, University of Heidelberg
Other Study IDs: TnT hs 4
Record Dates: First submitted 2011-04-13; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-03

CONDITIONS: Duration of Weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — routine blood parameters
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- weaning patients

SUMMARY:
The purpose of the study is to examine the relevance of biochemical markers (specific pulmonary and cardiac markers and markers of endogenous stress) in the process of weaning in patients with artificial ventilation.

DETAILED DESCRIPTION:
Artificially ventilated patients on our intensive care unit will be monitored if specific biomarkers have a relevance in risk stratification, optimizing therapy, outcome and success in the process of weaning. Therefore, consecutively, specific blood parameters will be taken at time of intubation,day 1 of weaning and extubation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Able and willing to understand the protocol
* At least 18 years or older

Exclusion Criteria:

* Not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutively all patients on our intensive care unit who are artificially ventilated
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
success of weaning | participants will be followed for the duration of hospital stay, an expected average of 30days
  primary outcome measure is the success of weaning during hospital stay. Duration of hospital stay is estimated between 1-60days, in average 30days. Criteria is spontaneous breathing.

SECONDARY OUTCOMES:
follow up | 12 months
  Follow up is done after 12 months to check major adverse cardiac or pulmonary events (death, myocardial infarction, re-hospitalisation)

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany